CLINICAL TRIAL: NCT01665924
Title: Single and Multiple Dose Pharmacokinetics of GLPG0634 in Elderly Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLPG0634-CL-104
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG0634

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 40-50 years old (Experimental): GLPG0634 100mg capsule once a day for 10 days in healthy subjects between 40 and 50 years old
  Interventions: Drug: GLPG0634 100mg capsule once a day for 10 days
- 65-74 years old (Experimental): GLPG0634 100mg capsule once a day for 10 days in healthy subjects between 65 and 74 years old
  Interventions: Drug: GLPG0634 100mg capsule once a day for 10 days
- 75 years and older (Experimental): GLPG0634 100mg capsule once a day for 10 days in healthy subjects of 75 years and older
  Interventions: Drug: GLPG0634 100mg capsule once a day for 10 days

INTERVENTIONS:
Drug: GLPG0634 100mg capsule once a day for 10 days

SUMMARY:
The purpose of the study is to evaluate the amount of compound present in the blood (pharmacokinetics) after single and of multiple doses of GLPG0634 in elderly healthy subjects.

During the course of the study, the effect of aging on the pharmacokinetics as well as the effects of GLPG0634 on mechanism of action-related parameters in the blood (pharmacodynamics) will be assessed and the safety of multiple oral doses of GLPG0634 in elderly healthy subjects will be characterized.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, age 40 years and older
* BMI between 18-30 kg/m2

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The amount of GLPG0634 in plasma over time after single and multiple doses of GLPG0634 | From predose (before first study drug administration) up to 72 hours post last study drug administration
  To characterize the amount of GLPG0634 in plasma over time - pharmacokinetics (PK) - after single and multiple oral doses in different age groups, including elderly healthy subjects, thereby assessing the effect of aging

SECONDARY OUTCOMES:
The amount of GLPG0634 mechanism-of-action-related biomarkers in blood after multiple doses of GLPG0634 | From predose (before first study drug administration) up to 24 hours post last study drug administration
  To characterize the effects of GLPG0634 on mechanism of action-related biomarkers in the blood over time - pharmacodynamics (PD) - after multiple oral doses in different age groups, including elderly healthy subjects, thereby assessing the effect of aging
Number of adverse events | From screening up to 10 days after the last study drug administration
  To evaluate the safety of multiple oral doses of GLPG0634 in healthy subjects of different age groups, including elderly, in terms of the number of adverse events reported
Changes in vital signs as measured by heart rate, blood pressure and body temperature | From screening up to 10 days after the last study drug administration
  To evaluate the safety of multiple oral doses of GLPG0634 in healthy subjects of different age groups, including elderly, in terms of changes in vital signs as measured by heart rate, blood pressure and body temperature reported
Changes in 12-lead ECG measures | From screening up to 10 days after the last study drug administration
  To evaluate the safety of multiple oral doses of GLPG0634 in healthy subjects of different age groups, including elderly, in terms of changes in 12-ECG measures reported
Changes in physical exam measures | From screening up to 10 days after the last study drug administration
  To evaluate the safety of multiple oral doses of GLPG0634 in healthy subjects of different age groups, including elderly, in terms of changes in physical examination reported
Changes in blood safety lab parameters | From screening up to 10 days after the last study drug administration
  To evaluate the safety of multiple oral doses of GLPG0634 in healthy subjects of different age groups, including elderly, in terms of changes in blood safety lab parameters assessed
Changes in urine safety lab parameters | From screening up to 10 days after the last study drug administration
  To evaluate the safety of multiple oral doses of GLPG0634 in healthy subjects of different age groups, including elderly, in terms of changes in urine safety lab parameters assessed

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV; Magdalena Petkova, MD, Principal Investigator — SGS LSS Clinical Pharmacology Unit Antwerp
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Antwerp, Belgium